CLINICAL TRIAL: NCT03796741
Title: STable Coronary Artery Diseases RegisTry
Acronym: START
Status: Completed | Type: Observational
Sponsor: Heart Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: K14
Record Dates: First submitted 2018-12-20; First posted 2019-01-08 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2018-12

CONDITIONS: Chronic Ischemic Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection on Stable Ischemic heart disease — No intervention only description of management and treatment

SUMMARY:
Observational, prospective multicentric, national study, evaluating the diagnostic and therapeutic pathways of patient with cronic coronary artery disease followed in Italian cardiology centers.

DETAILED DESCRIPTION:
Coronary heart disease is still highly prevalent in the world, and chronic stable angina is one of the most common clinical presentations of this disease. The objectives of chronic stable angina treatment include the reduction of symptoms, the inhibition or slowing of the progression of the disease, the prevention of associated cardiovascular events such as myocardial infarction, and the possible improvement of survival.The results of COURAGE Study and of meta-analysis of more recent studies demonstrate that patients in optimized medical therapy (OMT) (aspirin, beta-blocker and statin in association with an ACE-inhibitor and strict control of risk factors). ) the percutaneous coronary revascularization procedure (PCI) did not lead to an improvement in the cardiovascular prognosis. These data led the groups in charge of drafting the guidelines to recommend OMT as an initial treatment of stable angina, reserving the revascularization procedure for those patients with symptoms not adequately controlled by medical therapy.

It is therefore considered appropriate to plan a registry in patients with stable coronary artery disease that has the ability to describe in the heterogeneity of Italian cardiological centers the current characteristics of these patients, their treatment modalities, adherence to the current guidelines both as regards invasive therapy that the optimized medical, the use and the total cost of the resources needed to manage this pathology, the clinical course one year after entering the register.

Consecutive patients discharged (after an ordinary or day hospital admission) or managed as outpatient at Cardiology department participating in the project with a diagnosis of stable coronary artery disease will be included in the register. Enrollment will last 3 months in each center, starting with the first enrolled patient, or up to 50 patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >/= 18
* Patients discharged from hospital or ambulatory visit with a diagnoses of stable heart disease;
* Written informed consent

Exclusion Criteria:

* Acute coronary syndrome within 30 days from enrollment
* CCS Angina Class IV
* Angina probably not for coronary artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients discharged (after a hospitalization or DH hospitalization) or managed as outpatients in Cardiology department with diagnoses of stable coronary heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 5070 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Number of patients in medical therapy and that underwent revascularization | Enrollment
  Number of patients in medical therapy and that underwent revascularization

SECONDARY OUTCOMES:
Number of patient in optimal medical therapy | 12 months Follow-up
  Patient treated according to International Guidelines
Mortality rate | 12 months Follow-up
  Rate of patients died
All cause hospitalization rate | 12 months Follow-up
  Rate of patients hospitalized
Angina recurrence rate | 12 months Follow-up
  Rate of patients with angina symtoms

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo De Luca, MD, Study Chair — Heart Care Foundation
Locations (183):
- Italy (183):
  - Ospedale San Giovanni Di Dio - Uo Cardiologia E Utic, Agrigento, AG
  - Istituto Scientifico Inrca - Uo Cardiologia/Utic/Telecardiologia, Ancona, AN
  - Ospedale Civile Profili - U.O. Cardiologia, Fabriano, AN
  - Ospedale Di Jesi Carlo Urbani - U.O. Di Cardiologia, Iesi, AN
  - Ospedale Principe Di Piemonte - Uoc Cardiologia Utic, Senigallia, AN
  - Ospedale Gen.Le Prov.Le C.G. Mazzoni - Sc Cardiologia, Ascoli Piceno, AP
  - Ospedale Madonna Del Soccorso - Uoc Cardiologia Indirizzo Riabilitativo, San Benedetto del Tronto, AP
  - Ospedale Valdichiana Santa Margherita - Uos Cardiologia E Hdu, Cortona, AR
  - Aorn San Giuseppe Moscati - U.O. Cardiologia/Utic 'D. Rotiroti', Avellino, AV
  - Ospedale San Paolo - Cardiologia-Utic, Bari, BA
  - Ospedale Policlinico - U.O. Di Cardiologia Ospedaliera, Bari, BA
  - Ics Maugeri Spa Societa' Benefit - Uo Cardiologia, Cassano delle Murge, BA
  - Ospedale Umberto I - Uosd Di Cardiologia, Corato, BA
  - P.O. Don Tonino Bello - Uosd Cardiologia, Molfetta, BA
  - Asst Papa Giovanni Xxiii - Cardiologia 1, Bergamo, BG
  - Iob - Policlinico San Marco - U.O. Cardiologia, Osio Sotto, BG
  - Ospedale Civile - Sc Cardiologia, Belluno, BL
  - Ospedale Santa Maria Del Prato - U.O. Di Cardiologia, Feltre, BL
  - Azienda Ospedaliera G. Rummo - Cardiologia Interventistica E Utic, Benevento, BN
  - Ospedale Perrino - U.O.C. Di Cardiologia, Brindisi, BR
  - Ospedale Civile Dario Camberlingo - U.O. Di Cardiologia - Utic, Francavilla Fontana, BR
  - Ospedale Civile 'La Memoria' - U.O. Di Cardiologia, Gavardo, BS
  - Ics Maugeri Spa Societa' Benefit - U.O. Di Cardiologia Riabilitativa, Lumezzane, BS
  - Osp. Andria Canosa - Po Andria - Cardiologia - Utic, Andria, BT
  - Ospedale Monsignor Angelo R. Di Miccoli - Unita' Operativa Di Cardiologia, Barletta, BT
  - Presidio Ospedaliero Ss Trinita' - Sc Di Cardiologia, Cagliari, CA
  - Azienda Ospedaliera G. Brotzu - Struttura Complessa Di Cardiologia, Cagliari, CA
  - Ospedale A. Cardarelli - U.O. Cardiologia E Utic, Campobasso, CB
  - Presidio Ospedaliero Moscati - U.O.C. Cardiologia, Aversa, CE
  - Az. Ospedaliera S. Anna E S. Sebastiano - Cardiologia E Riabilit. Cardiologica, Caserta, CE
  - Az. Ospedaliera S. Anna E S. Sebastiano - U.O. Cardiologia-Utic, Caserta, CE
  - Pineta Grande Hospital - U.O. Cardiologia, Castel Volturno, CE
  - Ospedale Civile Ave Gratia Plena - U.O. Di Cardiologia E Utic, Piedimonte Matese, CE
  - Ospedale San Giuseppe E Melorio - U.O.C. Cardiologia Utic, Santa Maria Capua Vetere, CE
  - Presidio Ospedaliero San Rocco - U.O.C. Cardiologia - Utic, Sessa Aurunca, CE
  - Po Vittorio Emanuele Di Gela - U.O.C Cardiologia - Utic, Gela, CL
  - Ospedale Moriggia Pelascini - Unita' Operativa Di Cardiologia, Gravedona, CO
  - Ospedale Civile Oglio Po - U.O. Di Cardiologia-Utic, Casalmaggiore, CR
  - Ospedale Di Cremona - Uo Di Cardiologia, Cremona, CR
  - Capt Di Cariati - Ambulatorio Di Cardiologia, Cariati, CS
  - Ospedale Annunziata - Uoc Cardiologia, Cosenza, CS
  - Ospedale Civile Minervini - Medicina Interna, Mormanno, CS
  - P.O. Garibaldi-Nesima - U.O.C. Di Cardiologia, Catania, CT
  - Ospedale Giovanni Paolo Ii - U.O. Cardiologia E Utic, Lamezia Terme, CZ
  - I.R.C.C.S. Oasi Maria Ss. - U.O. Cardiologia, Troina, EN
  - Ospedale M.Bufalini - U.O. Di Cardiologia-Utic, Cesena, FC
  - Ospedale Ss. Annunziata - U.O. Di Cardiologia, Cento, FE
  - Arcispedale Sant'Anna - U.O. Cardiologia - Utic, Ferrara, FE
  - Ospedale Civile Giuseppe Tatarella - U.O. Di Cardiologia - Utic, Cerignola, FG
  - Ospedali Riuniti - S.C. Di Cardiologia Univ.-Utic, Foggia, FG
  - Ospedale Casa Sollievo Della Sofferenza - Cardiologia - Utic - Riabil Cardiologica, San Giovanni Rotondo, FG
  - Ospedale Civile Augusto Murri - U.O. Cardiologia, Fermo, FM
  - Ospedale Padre Antero Micone - Sc Cardiologia - Utic, Genova, GE
  - Ospedale San Giovanni Di Dio - S.O.C. Cardiologia, Gorizia, GO
  - Ospedale Civile San Polo - S.O.C. Cardiologia, Monfalcone, GO
  - Ospedale Della Misericordia - U.O. Di Cardiologia, Grosseto, GR
  - Ospedale Civile - U.O. Cardiologia-Utic, Imperia, IM
  - Presidio Ospedaliero - U.O. Cardiologia, Sanremo, IM
  - Ospedale F. Veneziale - Ssd Cardiologia Emodinamica, Isernia, IS
  - Ospedale San Giuseppe Da Copertino - U.O. Di Cardiologia-Utic, Copertino, LE
  - Ospedale Santa Caterina Novella - U.O. Di Cardiologia, Galatina, LE
  - Casa Di Cura Petrucciani - U.O. Cardiologia - Card. Riabilitativa, Lecce, LE
  - Ospedale Vito Fazzi - U.O. Card. Interventistica - Emodinamica, Lecce, LE
  - Ospedale Vito Fazzi - U.O. Di Cardiologia, Lecce, LE
  - Ospedale Ignazio Veris Delli Ponti - Uoc Cardiologia-Utic, Scorrano, LE
  - Azienda Osp. Cardinale G. Panico - U.O. Cardiologia - Utic, Tricase, LE
  - Ospedale Villamarina - Cardiologia E Utic, Piombino, LI
  - Casa Di Cura Citta' Di Aprilia - U.O. Cardiologia, Aprilia, LT
  - Ospedale Del Dono Svizzero - U.O.C. Di Cardiologia - Utic, Formia, LT
  - Polo Ospedaliero Integrato (C/O Icot) - Uoc Cardiologia Ed Emodinamica Univ., Latina, LT
  - Nuovo Ospedale Versilia - Sc Cardiologia, Lido di Camaiore, LU
  - Ospedale Carate Brianza - Cardiologia - Carate Brianza/Giussano, Carate Brianza, MB
  - Policlinico Di Monza - Uo Cardiol. Clinica E Scompenso Cardiaco, Monza, MB
  - Presidio Osp. Di Civitanova Marche - Sc Cardiologia, Civitanova Marche, MC
  - P.O. Sant'Agata Di Militello - Uoc Cardiologia, Sant'Agata di Militello, ME
  - Ospedale Civile - Uo Cardiologia, Legnano, MI
  - Ospedale Civile Fornaroli - U.O. Cardiologia, Magenta, MI
  - Istituto Clinico Citta' Studi - U.O. Cardiologia, Milan, MI
  - Ospedale San Raffaele - Utic E Subintensiva, Milan, MI
  - Ospedale San Carlo Borromeo - Cardiologia-Ucc, Milan, MI
  - Istituto Clinico Humanitas - Uo Emodinamica Cardiologia Invasiva Ucc, Rozzano, Mi
  - Irccs Policlinico San Donato - U.O. Cardiologia Con Utic, San Donato Milanese, MI
  - Irccs Policlinico Multimedica - Uo Di Cardiologia, Sesto San Giovanni, MI
  - Ospedale Di Vizzolo Predabissi - Uo Cardiologia E Ucc, Vizzolo Predabissi, MI
  - Ospedale Di Sassuolo - Cardiologia, Sassuolo, MO
  - Ftgm - Stabilimento Di Massa - Uoc Cardiologia Diagn. E Interventistica, Massa, MS
  - Ospedale Apuane - U.O. Cardiologia-Utic, Massa, MS
  - Ospedale San Francesco - Cardiologia - Utic, Nuoro, NU
  - Casa Di Cura Candela - Uof Cardiologia, Palermo, PA
  - Aor Villa Sofia-Cervello P.O. Cervello - U.O. Cardiologia - Cervello, Palermo, PA
  - Ospedale Di Camposampiero - U.O.A. Cardiologia, Camposampiero, PD
  - Ospedale Civile Dello Spirito Santo - Utic E Cardiologia Interventistica, Pescara, PE
  - Presidio Ospedaliero Citta' Di Castello - U.O. Di Cardiologia, Città di Castello, PG
  - Ospedale Di Pordenone - S.O.C. Cardiologia, Pordenone, PN
  - Ospedale Di S. Vito Al Tagliamento - S.O.C. Cardiologia, San Vito al Tagliamento, PN
  - Fondazione Irccs Policlinico San Matteo - Cardiologia, Pavia, PV
  - Ics Maugeri Spa Societa' Benefit - U.O. Di Riabilitazione Cardiologica, Pavia, PV
  - Istituto Di Cura Citta' Di Pavia - U.O. Cardiologia Ii, Pavia, PV
  - Ospedale Civile - Cardiologia, Vigevano, PV
  - Ospedale S. Giovanni Di Dio - U.O. Cardiologia E Utic, Melfi, PZ
  - Azienda Ospedaliera San Carlo - S.S.D. Cardiologia Riabilitativa, Potenza, PZ
  - Ospedale Per Gli Infermi - U.O. Cardiologia - Utic, Faenza, RA
  - Ospedale Civile - U.O. Di Cardiologia, Lugo, RA
  - Ospedale Civile Santa Maria Delle Croci - U.O. Di Cardiologia, Ravenna, RA
  - Ospedale Civile - S.O.C. Cardiologia-Utic, Locri, RC
  - Ospedale Tiberio Evoli Riabilitazione - Cardio-Respiratoria, Melito di Porto Salvo, RC
  - Ospedale Santa Maria Degli Ungheresi - U.O. Di Cardiologia, Polistena, RC
  - Ao Bianchi Melacrino Morelli- Po Riuniti - Divisione Di Cardiologia, Reggio Calabria, RC
  - Ospedale Civile San Sebastiano - Sos Cardiologia Area Nord, Correggio, RE
  - Ospedale Civile - Sc Cardiologia Area Nord, Guastalla, RE
  - Arcispedale Santa Maria Nuova - S.C. Cardiologia, Reggio Emilia, RE
  - Giovanni Paolo Ii - U.O.C. Cardiologia-Utic, Ragusa, RG
  - Ospedale Riccardo Guzzardi - U.O.C. Di Cardiologia-Utic, Vittoria, RG
  - P.O. San Camillo de Lellis - U.O.C. Cardiologia, Rieti, RI
  - Ospedali Riuniti Anzio-Nettuno - U.O. Di Cardiologia - Utic, Anzio, RM
  - Nuovo Ospedale Dei Castelli - U.O.C. Di Cardiologia E Utic, Ariccia, RM
  - Ospedale Civile San Paolo - U.O. Cardiologia - Utic, Civitavecchia, RM
  - Policlinico Citta' Di Pomezia S. Anna - U.O. Cardiologia-Utic, Pomezia, RM
  - Campus Biomedico - Cardiologia, Roma, RM
  - P.O. San Filippo Neri - Asl Roma 1 - Uoc Cardiologia E Utic, Roma, RM
  - European Hospital - Uo. Cardiologia Interventistica, Roma, RM
  - Ospedale San Camillo - Cardiologia 2 (Ex Cardio 3), Roma, RM
  - Ospedale San Camillo - Uoc Cardiologia 1, Roma, RM
  - Ospedale Sandro Pertini - Uoc Cardiologia, Roma, RM
  - Policlinico Umberto Primo - Cardiologia B - Cardiologia E Angiologia, Roma, RM
  - Policlinico Umberto Primo - Malattie Cardiovascolari A, Roma, RM
  - Aurelia Hospital - U.O.C Cardiologia, Roma, RM
  - Ospedale Madre Giuseppina Vannini - U.O.C. Cardiologia, Roma, RM
  - Ospedale San Pietro Fatebenefratelli - U.O Complessa Di Cardiologia, Roma, RM
  - Ospedale Sant'Andrea Di Roma - U.O.C. Cardiologia, Roma, RM
  - Ospedale Santo Spirito - U.O.C. Di Cardiologia, Roma, RM
  - Ospedale San Giovanni Evangelista - U.O.C. Di Cardiologia - Utic, Tivoli, RM
  - Ospedale Santa Maria Della Misericordia - U.O.C. Cardiologia, Rovigo, RO
  - Presidio Osped. S. Maria Della Speranza - U.O. Di Cardiologia, Battipaglia, SA
  - Ospedale Di Roccadaspide - Cardiologia-Utic, Roccadaspide, SA
  - Aou S. Giovanni Di Dio-Ruggi D'Aragona - Uoc Cardiologia Preventiva, Salerno, SA
  - Ospedale San Luca - U.O. Utic - Cardiologia, Vallo della Lucania, SA
  - Ospedale Dell'Alta Val D'Elsa - Uosd Cardiologia-Utic, Poggibonsi, SI
  - Aou Senese Ospedale S. Maria Alle Scotte - U.O.C. Cardiologia Ospedaliera, Siena, SI
  - Ospedale San Bartolomeo - U.O. Cardiologia Clinica-Riabilitativa, Sarzana, SP
  - Ospedale E. Muscatello - U.O. Di Cardiologia - Utic, Augusta, SR
  - Ospedale G. Di Maria - Cardiologia Utic, Avola, SR
  - Ospedale Umberto I - Uoc Cardiologia E Utic, Syracuse, SR
  - Ospedale Civile M. Giannuzzi - Cardiologia E Utic, Manduria, TA
  - Casa Di Cura Villa Verde - Cardiologia, Taranto, TA
  - Ospedale Civile G. Mazzini -Cardiologia Utic Ed Emodinamica, Teramo, TE
  - Ospedale Santa Chiara - Divisione Di Cardiologia, Trento, TN
  - Por Cirie'- Lanzo Presidio Cirie' - S.C. Cardiologia Cirie'- Ivrea, Cirié, TO
  - Ospedale Civile - S.C. Cardiologia Cirie' Ivrea, Ivrea, TO
  - Maria Pia Hospital - U.O. Cardiologia, Torino, TO
  - Ospedale Ss. Vito E Spirito - U.O.S. Di Cardiologia, Alcamo, TP
  - Presidio Ospedaliero Paolo Borsellino - U.O.C Cardiologia- Utic, Marsala, TP
  - Ospedale S. Maria Della Stella - Sc Di Cardiologia, Orvieto, TR
  - Ospedali Riuniti - Osp. Maggiore - A.F. Cardiologia E Riabil. Cardiologica, Trieste, TS
  - Ospedale Santa Maria Dei Battuti - U.O. Di Cardiologia, Conegliano, TV
  - Pou Santa Maria Della Misericordia - S.O.C. Cardiologia, Udine, UD
  - Ospedale S. Antonio Abate - U.O. Di Cardiologia, Gallarate, VA
  - Presidio Ospedaliero Di Saronno - U.O.C. Di Cardiologia, Saronno, VA
  - Ospedale Di Circolo A. Bellini - Medicina Generale E Card. Riabilitativa, Somma Lombardo, VA
  - Ospedale Di Circolo Galmarini - Cardiologia, Tradate, VA
  - Ospedale Di Circolo E Fondazione Macchi - Cardiologia I, Varese, VA
  - Ospedale Sant'Andrea - Sc Cardiologia, Vercelli, VC
  - Ospedale Civile - U.O.C. Cardiologia, Chioggia, VE
  - Ospedale Civile Di Venezia - U.O. Di Cardiologia, Venezia, VE
  - Ospedale Civile - U.O.C. Cardiologia, Arzignano, VI
  - Centro Polifunzionale Boldrini - Cardiologia Riabilitativa-Cardioaction, Thiene, VI
  - Ospedale G. Fracastoro - U.O.C. Di Cardiologia, San Bonifacio, VR
  - Ospedale Belcolle - U.O.C. Cardiologia Utic Emodinamica, Viterbo, VT
  - Clinica Citta' Di Alessandria - Uo Cardiologia, Alessandria
  - Ospedale Civile Di Boscotrecase - Utic Cardiologia, Boscotrecase
  - Ospedale San Giovanni Di Dio - Uo Cardiologia - Utic, Frattamaggiore
  - Ospedale Generale Di Zona - U.O. Cardiologia - Utic, Giugliano in Campania
  - Clinica Mediterranea - U.O. Di Cardiologia, Napoli
  - Aorn Cardarelli - U.O. Cardiologia Con Utic, Napoli
  - Aorn Osp. Dei Colli- Po Vincenzo Monaldi - U.O.C. Cardiologia E Utic 'Vanvitelli', Napoli
  - Aorn Osp. Dei Colli- Po Vincenzo Monaldi - U.O.C. Cardiologia, Napoli
  - Ospedale San Gennaro - U.O. Cardiologia E Riabilitazione Card., Napoli
  - Ospedale Del Mare - U.O. Cardiologia Con Utic, Napoli
  - Aou Maggiore Della Carita' - Cardiologia Ii, Novara
  - Aou Maggiore Della Carita' Scdu Clinica Cardiologica-Cardiologia I, Novara
  - Clinica San Gaudenzio - Uoa Cardiologia, Novara
  - Casa Di Salute Santa Lucia - U.O. Cardiologia, San Giuseppe Vesuviano
  - Ics Maugeri Spa Societa' Benefit - Uo Cardiologia Riabilitativa, Veruno

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Luca L, Temporelli PL, Lucci D, Colivicchi F, Calabro P, Riccio C, Amico A, Mascia F, Proia E, Di Lenarda A, Gulizia MM; START Investigators. Characteristics, treatment and quality of life of stable coronary artery disease patients with or without angina: Insights from the START study. PLoS One. 2018 Jul 12;13(7):e0199770. doi: 10.1371/journal.pone.0199770. eCollection 2018. PMID 30001355
- [Background] De Luca L, Arca M, Temporelli PL, Colivicchi F, Gonzini L, Lucci D, Bosco B, Callerame M, Lettica GV, Di Lenarda A, Gulizia MM; START Investigators. Prevalence and pharmacologic management of familial hypercholesterolemia in an unselected contemporary cohort of patients with stable coronary artery disease. Clin Cardiol. 2018 Aug;41(8):1075-1083. doi: 10.1002/clc.23031. Epub 2018 Aug 20. PMID 30039543
- [Background] Colivicchi F, Massimo Gulizia M, Arca M, Luigi Temporelli P, Gonzini L, Venturelli V, Morici N, Indolfi C, Gabrielli D, De Luca L. Lipid Lowering Treatment and Eligibility for PCSK9 Inhibition in Post-Myocardial Infarction Patients in Italy: Insights from Two Contemporary Nationwide Registries. Cardiovasc Ther. 2020 Jan 3;2020:3856242. doi: 10.1155/2020/3856242. eCollection 2020. PMID 31969932
- [Background] De Luca L, Arca M, Temporelli PL, Meessen J, Riccio C, Bonomo P, Colavita AR, Gabrielli D, Gulizia MM, Colivicchi F; START Investigators. Current lipid lowering treatment and attainment of LDL targets recommended by ESC/EAS guidelines in very high-risk patients with established atherosclerotic cardiovascular disease: Insights from the START registry. Int J Cardiol. 2020 Oct 1;316:229-235. doi: 10.1016/j.ijcard.2020.05.055. Epub 2020 May 26. PMID 32470532
- [Background] De Luca L, Formigli D, Meessen J, Uguccioni M, Cosentino N, Paolillo C, Di Lenarda A, Colivicchi F, Gabrielli D, Gulizia MM, Scherillo M; START Investigators. COMPASS criteria applied to a contemporary cohort of unselected patients with stable coronary artery diseases: insights from the START registry. Eur Heart J Qual Care Clin Outcomes. 2021 Sep 16;7(5):513-520. doi: 10.1093/ehjqcco/qcaa054. PMID 32559279
- [Background] De Luca L, Uguccioni M, Meessen J, Temporelli PL, Tomai F, De Rosa FM, Passamonti E, Formigli D, Riccio C, Gabrielli D, Colivicchi F, Gulizia MM, Perna GP. External applicability of the ISCHEMIA trial: an analysis of a prospective, nationwide registry of patients with stable coronary artery disease. EuroIntervention. 2020 Dec 18;16(12):e966-e973. doi: 10.4244/EIJ-D-20-00610. PMID 32830646
- [Background] De Luca L, Temporelli PL, Amico AF, Gonzini L, Uguccioni M, Varani E, Brunetti ND, Colivicchi F, Gabrielli D, Gulizia MM. Impact of history of depression on 1-year outcomes in patients with chronic coronary syndromes: An analysis of a contemporary, prospective, nationwide registry. Int J Cardiol. 2021 May 15;331:273-280. doi: 10.1016/j.ijcard.2020.12.086. Epub 2021 Jan 8. PMID 33422564
- [Result] De Luca L, Temporelli PL, Lucci D, Gonzini L, Riccio C, Colivicchi F, Geraci G, Formigli D, Maras P, Falcone C, Di Lenarda A, Gulizia MM; START Investigators. Current management and treatment of patients with stable coronary artery diseases presenting to cardiologists in different clinical contexts: A prospective, observational, nationwide study. Eur J Prev Cardiol. 2018 Jan;25(1):43-53. doi: 10.1177/2047487317740663. Epub 2017 Nov 10. PMID 29124952
- [Result] De Luca L, Temporelli PL, Riccio C, Gonzini L, Marinacci L, Tartaglione SN, Costa P, Scherillo M, Senni M, Colivicchi F, Gulizia MM; START Investigators. Clinical outcomes, pharmacological treatment, and quality of life of patients with stable coronary artery diseases managed by cardiologists: 1-year results of the START study. Eur Heart J Qual Care Clin Outcomes. 2019 Oct 1;5(4):334-342. doi: 10.1093/ehjqcco/qcz002. PMID 30649303